CLINICAL TRIAL: NCT06938542
Title: Palliative Care Needs of Children With Rare Diseases and Their Families
Acronym: FACE-Rare
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Children's National Research Institute (Other)
Collaborators: Akron Children's Hospital (Other); Stanford University (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Maureen Lyon, Clinical Psychologist, Tenured Professor of Pediatrics, Children's National Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: R01HD117137-01 (NIH); 1R01HD117137-01 (NIH)
Record Dates: First submitted 2025-04-08; First posted 2025-04-22 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Trisomy 13 Syndrome; Arthrogryposis Congenita Multiplex With Intestinal Atresia; Asparagine Synthetase Deficiency; CHARGE Syndrome; Early Infantile Epileptic Encephalopathy; FOXG1 Syndrome; KBG Syndrome; Noonan Syndrome; Severe Hemophilia A; Short Bowel Syndrome; Beta-Propeller Protein-Associated Neurodegeneration; Brain Injury of Prematurity With Periventricular Leukomalacia; Chromosome 17p13.3 Microdeletion Syndrome; Chromosome 1q43-1q44 Deletion; Cockayne Syndrome; Congenital Diaphragmatic Hernia; End-Stage Renal Disease With Cloacal Anomaly; Mitochondrial Depletion Disorder; Severe Factor VII Deficiency
Keywords: pediatrics; palliative care; rare diseases; rare disorders; randomized clinical trial; advance care planning; quality of life; social connection; intervention; spirituality; anxiety; depression; caregiving
MeSH Terms: conditions — Trisomy 13 Syndrome; CHARGE Syndrome; Infantile Epileptic-Dyskinetic Encephalopathy; KBG syndrome; Noonan Syndrome; Hemophilia A; Short Bowel Syndrome; Cockayne Syndrome; Hernias, Diaphragmatic, Congenital; Factor VII Deficiency; Rare Diseases; Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FACE-Rare (Experimental): FACE-Rare (CSNAT-P Sessions 1 & 2 plus Next Steps: Respecting Choices Sessions 3). The CSNAT-Pediatric intervention consists of two assessment visits with the facilitator, 2-8 weeks apart, comprising conversations about sources for support in a tertiary children's hospital. The adapted Next Steps: Respecting Choices pediatric Advance Care Planning conversation engages families in a process for how to make future medical decisions consistent with the families' goals and values. The Respecting Choices structured and facilitated conversation has five stages. Stage 1: Assesses the family's understanding of illness. Stage 2: Explores experiences with hospitalization. Stage 3: Explores goals of care. Stage 4: Creates an Advance Care Plan; Stage 5: Questions for providers are written down. Stage 6: Follow-up plan and referrals, as needed.
  Interventions: Behavioral: Family Centered pediatric palliative care for family caregivers of children with rare diseases.
- Enhanced Treatment As Usual (TAU) (Experimental): Treatment as Usual Control (TAU): To minimize the burden to families, we have chosen an enhanced (palliative care information and resources) TAU comparison condition.
  Interventions: Behavioral: Family Centered pediatric palliative care for family caregivers of children with rare diseases.

INTERVENTIONS:
Behavioral: Family Centered pediatric palliative care for family caregivers of children with rare diseases. — Child with rare disease who is unable to participate in medical decision making/family caregiver/support person triads will be randomized at a 1:1 ratio to one of two study arms, either the 3 session FACE-Rare intervention or the enhanced Treatment as Usual. Assessments will be completed at baseline, 3, 6 and 12 month outcomes.

SUMMARY:
The palliative care needs of family caregivers of children with rare diseases and their children are largely unmet, including the need for support to prepare for future medical decision making. This trial will test the FACE-Rare intervention to see if investigators can identify and meet those needs; and if FACE-Rare effects family caregivers' quality of life and child healthcare utilization. Finally, investigators will determine if the intersectionality of child-sex, family-race, Federal poverty level, and social connection influences family quality of life and child health care utilization longitudinally.

DETAILED DESCRIPTION:
Pediatric patients with rare diseases experience high mortality with 30% not living to see their 5th birthday. Families are likely to be asked to make complex medical decisions for their child. Pediatric advance care planning involves preparation and skill development to help make future medical care choices. Children with rare disorders are a heterogeneous group, resulting in their exclusion from research. Available research on families of children with rare diseases lacks scientific rigor. Although desperately needed, there are few empirically validated interventions to address these issues. Investigators propose to close a gap in our knowledge of families' needs for support in a heterogeneous group of children with rare diseases; and to test an advance care planning intervention. The FAmily CEntered (FACE) pediatric advance care planning intervention is adapted to families with children who have rare diseases. Theoretically informed and developed and adapted by the principal investigator and key stakeholders, the proposed intervention will use Respecting Choices Next Steps Pediatric ACP™ for families whose child is unable to participate in health care decision-making. Our consultation with families of children with rare disorders and the National Organization for Rare Disorders (NORD) revealed that basic palliative care needs should be addressed first, prior to an advance care planning intervention. For the study to be able to meet this request, all families randomized to the intervention will first complete the Carer Support Needs Assessment Tool (CSNAT)© adapted by investigators for use in pediatrics. In the CSNAT Approach, facilitators assess caregivers' prioritized palliative care needs and develop Shared Action Plans for increasing informal social support. Thus, investigators propose an innovative 3-session FACE-Rare intervention, integrating two evidence-based approaches. Investigators will evaluate FACE-Rare using a scientifically rigorous intent-to-treat, assessor-blinded, longitudinal, prospective, three-site, randomized controlled trial design. Family/child triads (N=160) will be randomized to FACE-Rare (CSNAT Sessions 1 & 2 plus Respecting Choices Sessions 3) or an enhanced information Treatment as Usual control group. All families will complete questionnaires at baseline and follow-up at 3-, 6- and 12 months. Investigators will evaluate the effect of FACE-Rare on family quality of life (caregiver appraisal, psychological, spiritual). Investigators will assess the palliative care needs of families at four time points. Investigators will determine the intersectionality of child-sex, family-race, and household income on family caregiver quality of life and child healthcare utilization. Investigators will explore the influence of urban vs. rural setting and religious coping on quality-of-life outcomes. Investigators will use advanced statistical methods informed by statistical advice from rare disease investigators for clinical trials in small populations.

ELIGIBILITY:
Child inclusion criteria:

* ≥1.0 years and <18.0 years at enrollment.
* Unable to participate in end-of-life care decision-making.
* Has a rare disease as operationally defined by NIH's Genetic and Rare Diseases Information Center (GARD).
* Not under a Do Not Resuscitate Order or Allow a Natural Death Order.
* Not in the Intensive Care Unit.

Family caregiver inclusion criteria:

* > 18.0 years at enrollment.
* Child's family caregiver/legal guardian.
* Not known to be developmentally delayed.

Support person inclusion criteria:

* > 18.0 years at enrollment.
* Chosen by family caregiver.
* Not known to be developmentally delayed.

Exclusion Criteria:

* Family caregiver or support person is actively homicidal, suicidal, or psychotic at the time of enrollment.

Ages: 12 Months to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2025-10-02 (Actual); Primary Completion 2029-02-02 (Estimated); Study Completion 2029-08-02 (Estimated)

PRIMARY OUTCOMES:
Family Appraisal of Caregiving for Palliative Care (FACQ-PC) | Baseline, 3-, 6-, and 12 month post-intervention
  The FACQ-PC is a 25-item measure consists of four theoretically derived subscales: (i) caregiver strain, (ii) positive caregiving appraisals, (iii) caregiver distress, and (iv) family well-being. Scores are from 5 = strongly agree to 1 = strongly disagree. Investigators will not calculate a Total score. On the subscale scores for positive caregiving appraisals and family well-being, higher scores mean better outcomes, i.e. greater positive caregiving appraisals or family well-being. On the subscale scores for caregiver strain and caregiver distress, higher scores mean worse outcomes, i.e. greater caregiver strain or caregiver distress. The FACQ-PC subscale scores will be computed by taking the mean of the items (score range 1-5). Some items are reverse scored, depending on how the item is phrased, so that higher scores = higher amount of the subscale being measured. So the minimum value for each subscale is 1 and the maximum value for each subscale is 5.
Functional Assessment of Chronic Illness Therapy-Spirituality-12 Version 4 Expanded (FACIT-Sp-EX) | Baseline, 3-, 6-, and 12 month post-intervention
  Assessed construct of spiritual well-being. Two subscales Meaning/Peace (7 items) and Faith (5 items) and Total score (12 items) were calculated. on a 5-point Likert scale from 0=not at all to 5=very much. Some items are reverse scored. See www.facit.org Meaning/Peace subscale score range from minimum value of 0 to maximum value of 32. Higher scores indicate better meaning/peace.
  Faith subscale score range from 0 minimum value to maximum value of 16. Higher scores indicate better meaning/peace.
  Total score range is from 0 minimum value to maximum value of 92. Higher scores indicate better spiritual well-being.
Advance Care Plan for Child with Rare Disease Located in the Electronic Health Record (EHR). | Baseline and 1 year
  Documentation of an advance care plan for child with rare disease in the Electronic Health Record and decisional preference - to continue all treatments, to continue all treatments with exceptions noted, to provide comfort care only.
Child Healthcare Utilization: initiation of palliative care consultations | Baseline, 3-, 6-, 12-month.
  Using a standardized data abstraction form to count initiation of palliative care consultations during the study.
Generalized Anxiety Disorder-7 (GAD-7) | Baseline, 3-, 6-, 12-month
  Quality of life indicator with respect to emotional health-anxiety symptoms. 7 items. Higher scores indicate greater anxiety.
Patient Health Questionaire-9 (PHQ-9) | Baseline, 3-, 6-, 12-month
  Quality of life indicator with respect to emotional health-depressive symptoms. 9 items. Higer scores indicate higher symptoms of depression. A yes response to question 9 (self-harm) will trigger a referral.
Child Healthcare Utilization: # of days in palliative care before death. | Baseline, 3-, 6-, 12-month
  Using a standardized data abstraction form to count # of days in palliative care before death.
Child Healthcare Utilization: # of hospitalizations during study participation | Baseline, 3-, 6-, 12-month
  Using a standardized data abstraction form to count # of days hospitalized during the study.
Child Healthcare Utilization: # of Emergency Department visits during study participation | Baseline, 3-, 6-, 12-month
  Using a standardized data abstraction form to count # of days used Emergency Department during study.
Child Healthcare Utilization: # of days in the Intensive Care Unit (ICU) | Baseline, 3-, 6-, 12-month
  Using a standardized data abstraction form to count # of days was admitted to ICU during the study.
Child Healthcare Utilization: # of surgeries | Baseline, 3-, 6-, 12-month
  Using a standardized data abstraction form to count # of surgeries during the study.

OTHER OUTCOMES:
Demographic Questionnaire | Baseline
  Age of family caregiver, support person, and child.
Process Measure: Satisfaction Questionnaire | Week 4
  Study specific process measure to assess adverse events and benefit/burden of participation. 13 items. Higher scores indicate greater satisfaction. Items are on a 5-point Likert scale from strongly disagree to strongly agree. 6 items were negative (felt afraid, too much to handle, harmful, angry, sad, hurtful) and 7 items were positive (useful, helpful, load off my mind, satisfied, something I needed to do, courageous, worthwhile). Each subscale is scored separately. Higher score for positive scale was better outcome. Higher score for negative scale was worse outcome.
Process Measure: Role Stress | Baseline, 3-, 6-, 12-month
  Visual analogue scale 0-100. "How stressful is it for you to make medical decisions for your child?" 1 item.
Brief-Multidimensional Measure of Spirituality and Religion (Brief MMRS) | Baseline, 3-, 6-, 12-month
  Responses to 5 items from our previous research will be used to test moderator effects: "How often do you go to religious services? How often do you feel God's presence? how often do you pray privately? Do you identify as a religious person? Do you identify as a spiritual person?" Responses are on a 5 point likert scale. Higher scores indicated greater attendance at religious services, etc.
BRICS (Brazil, Russia, India, China, South Africa) National Institute of Nursing Research (NINR) Social Determinants of Health (SDOH) | Baseline, 3-, 6-, 12-month
  NINR/National Institute of Health: "The SDOH are the conditions in which people are born, grow, live, work and age…." 32 items. Social connection score (how often, talk on telephone with family, friends, neighbors; get together; attend church or religious services; belong to clubs or organizations; marital partner status) and 2023 Federal Poverty Level for household income. Health insurance and housing insecurity will be used in secondary analysis.
Health Resources and Services Administration (HRSA) Rural Health Grants Eligibility Analyzer | Baseline, 3-, 6-, 12-month
  Urban vs. rural setting. Address of participant is entered into the online analyzer, and it determines if this is a rural or urban setting which will be recorded in the data base.
Carer Alert Thermometer (CAT) | Sessions 1 and 2 -- 2 and 3-4 weeks post baseline
  Measures child and family caregiver palliative care needs: The CAT is an evidence-based, comprehensive tool comprising 12 questions (broad areas of support need), used to identify two domains of unmet support needs, the current caring situation and the health and well-being of the caregiver. There is a traffic light scoring system so caregivers can rate their support need as green (low), amber (medium), and red (high) indicating level of need and potential risk each alert poses to the caregiving situation. Administered only to intervention participants.
Demographic Questionnaire - Sex | Baseline.
  Sex of child, family caregiver and support person.
Demographic Questionnaire - Race | Baseline.
  Race of child, family caregiver, and support person
Demographic Questionnaire - Ethnicity | Baseline.
  Ethnicity of child, family caregiver, and support person.
Demographic Questionnaire - Marital status. | Baseline.
  Marital status of family caregiver and support person.
Demographic Questionnaire - Education. | Baseline.
  Education of family caregiver and support person.
Demographic Questionnaire - Federal Poverty Level. | Baseline.
  Income above or below the 2025 Federal Poverty Level. Number of persons living in the household and household income will be collected to calculate these data.

CONTACTS AND LOCATIONS:
Overall Officials: Maureen E Lyon, PhD, Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Hospital, Washington D.C., District of Columbia, United States